CLINICAL TRIAL: NCT01491867
Title: Evaluation of Continuous IOP Measurement and the Influence of Drug Induced IOP Decrease on the Measurement
Brief Title: Continuous Intraocular Pressure (IOP) Measurement and Ability to Detect Treatment Effect
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Semmelweis University (Other)
Responsible Party: Principal Investigator, Gabor Hollo, Principle Investigator, Semmelweis University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 4481/2011
Record Dates: First submitted 2011-12-12; First posted 2011-12-14 (Estimated); Last update posted 2013-03-22 (Estimated); Status verified 2013-03

CONDITIONS: Glaucoma; Ocular Hypertension
Keywords: intraocular pressure
MeSH Terms: conditions — Glaucoma; Ocular Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Travoprost arm (Experimental): All individuals receive travoprost 0.003% 1/day in both eyes after 6 weeks wash-out for 3 months
  Interventions: Drug: travoprost 0.003%

INTERVENTIONS:
Drug: travoprost 0.003% — Instillation of travoprost 0.003% 1/die in both eyes for 3 months

SUMMARY:
Continuous intraocular pressure (IOP) measurement with a contact lens sensor may provide more information on the drug-related IOP change than 24-hour IOP measurement with Goldmann applanation tonometry (GAT.

DETAILED DESCRIPTION:
* Participants are washed ot from all glaucoma medication for 6 weeks
* one eye per participant is investigated (study eye)
* 24-h intraocular pressure (IOP) curve is obtained with Goldmann tonometry and Sensimed contact lens sensor tonometry twice, in 14 days
* for Sensimed contact lens curves median values (in arbitrary units), for Goldmann applanation tonometry, mean and SD values are used to characterize the curves, for comparisions % changes are used for the corresponding time periods
* treatment (travoprost 0.005% 1/day) is given to all eyes for 3 months 24-h Goldmann and Sensimed IOP curves are repeated
* IOP curves are determined in arbitrary units and mmHg, respectively, and compared for reproducibility (untreated phase) and relative (%)change (untreated curve vs. under treatment curve) with both methods, respectively

ELIGIBILITY:
Inclusion Criteria:

* primary open-angle glaucoma (POAG), ocular hypertension(OHT)
* 18 years or older
* C/D <= 0.7
* no risk for visual field damage
* IOP > 22 mmHg

Exclusion Criteria:

* Pregnancy and lactation
* Known intolerance to travoprost, topical anesthetic
* Previous ocular surgery at any time
* Previous ocular laser treatment within 1 year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2011-12; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Continuous intraocular pressure (IOP) measurement | 3 months
  24-h intraocular pressure (IOP) decrease induced by travoprost 0.003% 1/day as measured with Goldmann tonometry and Sensimed contact lens sensor

SECONDARY OUTCOMES:
Continuous intraocula pressure (IOP) Measurement | 3 months
  Reproducibility of intraocular pressure measurements with the Sensimed contact lens sensor methods

CONTACTS AND LOCATIONS:
Overall Officials: Gabor Hollo, MD, Principal Investigator — Semmelweis University
Locations (2):
- Hungary (2):
  - Departement of Ophthalmology, Budapest, Pest County
  - Semmelweis University, Budapest